CLINICAL TRIAL: NCT05190042
Title: Clinical Study on Continuous Suture of Mucosal Defects After Endoscopic Mucosal Lesion Resection
Brief Title: Clinical Study on Continuous Suture of Endoscopic Mucosal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 307-GIE-Suture
Record Dates: First submitted 2021-11-23; First posted 2022-01-13 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Colonic Polyp; Gastrointestinal Neoplasms
Keywords: Endoscopic mucosal resection; Endoscopic submucosal dissection; Gastrolintestinal polyps; Continuous suture; Clips
MeSH Terms: conditions — Colonic Polyps; Gastrointestinal Neoplasms | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Masking Description: This was a single-blind study where patients were not informed about their randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous suture group (Experimental): Surgical sutures were used to completely close the post-EMR/ESD mucosal/submucosal defects.
  This group was set as a experimental group.
  Interventions: Device: Cotinuous suture
- Clips group (Active Comparator): Clips were used to completely close the post-EMR/ESD mucosal/submucosal defects. This group was set as a control group.
  Interventions: Device: Clips

INTERVENTIONS:
Device: Cotinuous suture — Cotinuous suture using surgery thread
  Arms: Continuous suture group
Device: Clips — Hemostatic clips
  Arms: Clips group

SUMMARY:
The use of clips to completely clip mucosal defects after ESD/EMR can reduce postoperative adverse events, but the rate of incomplete mucosal defects closure is high. The continuous suture technique can completely close the mucosal defects by using surgical sutures and clips to suture the mucosal defects after ESD/EMR. In this study, a clinical randomized controlled study was conducted in our hospital. A total of 62 enrolled patients were divided into two groups, 31 patients were set as a treatment group using continuous suture technique to close post-EMR/ESD mucosal/submucosal defects, the rest patients were set as a control group using clips. The safety and effectiveness of continuous sutures and clips to clamp the post-EMR/ESD mucosal/submucosal defect were compared in the two groups. The complete mucosal/submucosa defects closure rates were the primary outcome.

DETAILED DESCRIPTION:
Endoscopic submucosal resection (EMR) or submucosal dissection (ESD) for gastrointestinal lesions were used to treat early gastrointestinal cancer or large benign polyps, and their complete resection rates were high, which greatly reduce unnecessary surgical operations. However, after endoscopic resection of mucosal/submucosal lesions, large mucosal/submucosal defects may be created. These defects may cause more delayed postoperative adverse events (bleeding, perforation). The use of clips to completely seal the mucosal defect after gastrointestinal mucosal/submucosal lesion resection can significantly reduce postoperative adverse events, but the rate of incomplete mucosal defects closure is high. The surgical sutures combined with clips to close the mucosal defect after surgery significantly increased the complete closure rates of the post-EMR/ESD mucosal/submucosal defect. This study intends to further determine its safety and effectiveness through a clinical randomized controlled study, and standardize indications and contraindications. A total of 62 enrolled patients were allocated into two groups, 31 patients were set as a treatment group using continuous suture technique to close post-EMR/ESD mucosal/submucosal defects, the rest patients were set as a control group using clips. The safety and effectiveness of continuous sutures and clips to clamp the post-EMR/ESD mucosal/submucosal defect were compared in the two groups. The primary outcome was complete mucosal/submucosa defects closure rates. The secondary outcomes were the closure time, closure speed, and immediate bleeding during the operation as well as delayed bleeding, delayed perforation, and polyps syndrome after resection.

ELIGIBILITY:
Inclusion Criteria:

1. The indications for endoscopic resection were large (≥20mm in diameter), nonpedunculated, benign, and early malignant mucosal or submucosal gastric or colorectal lesions.
2. Written informed consent

Exclusion Criteria:

1. The tumor has spread to the muscularis layer, lymph nodes, or distal metastases;
2. Multiple lesions (≥20mm in diameter) ;
3. Underlying bleeding disorder;
4. The platelet count less than 50×10^9/L;
5. Serious cardio-pulmonary, hepatic or renal disease;
6. Intolerance to endoscopy;
7. Other high-risk conditions or disease (such as massive ascites, etc.);
8. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
The rates of complete closure of mucosal/submucosal defects | 1day
  When the clips were applied next to each other and there were no substantial submucosal areas in the closure line

SECONDARY OUTCOMES:
The duration time of closure | 1 day
  The duration of closure was defined as the interval from insertion of the first clip until complete or incomplete closure
The closure speed | 1day
  The closure speed was defined as the resection area divided by 10x the duration of the ligation procedure (cm2 /10 minutes).
Immediate bleeding | 1 day
  Immediate bleeding refers to those episodes of hemorrhage that occurred during the procedure and lasted more than 30 seconds or required endoscopic treatment.
Delayed bleeding | 14 days
  Delayed bleeding was defined as bleeding requiring emergency endoscopic hemostasis or transfusion or the presence of hemoglobin loss≥2 g/dL after EMR/ESD
Delayed perforation | 14 days
  Delayed perforation was defined as the presence of free air on abdominal CT or radiography after completion of the procedure in patients without perforation during EMR/ESD and no symptoms of peritoneal irritation after EMR/ESD
Post polypectomy syndrome | 14 days
  Post polypectomy syndrome was defined by symptoms of pain, fever, leukocytosis, peritoneal tenderness, and guarding.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No